CLINICAL TRIAL: NCT04664101
Title: REmotely Monitored, Mobile Health-Supported High Intensity Interval Training After COVID-19 Critical Illness (REMM-HIIT-COVID-19)
Acronym: REMMHIIT-COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Vanderbilt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00105798
Record Dates: First submitted 2020-12-10; First posted 2020-12-11 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Covid19; Critical Illness; High Intensity Interval Training; ICU; Intensive Care Units; Fitness Trackers
Keywords: critical care; Covid19; ICU; high intensity interval training; intensive care unit; critical illness; fitness trackers
MeSH Terms: conditions — COVID-19; Critical Illness | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REmotely Monitored, Mhealth (REMM) supported High Intensity Interval Training (HIIT) (Experimental): REmotely Monitored, Mhealth (REMM) supported High Intensity Interval Training (HIIT) The intervention consists of high intensity interval training, consisting of a 30-minute exercise session that includes 10 x 1-minute intervals of high intensity 3x/week (e.g., Monday, Wednesday, Friday) and supplemented with 2 sessions per week of strength, balance, and mobility exercises (e.g., Tuesday, Thursday). Exercise will be supported by an activity tracker, which will allow study personnel to track patient heart rates during exercise on a daily basis, allowing them to provide individualized feedback and coaching.
  Interventions: Behavioral: REmotely Monitored, Mhealth (REMM) supported High Intensity Interval Training (HIIT)
- Comparator (Other): Patients randomized to the control arm will receive the same technology platform and education on exercise options, including HIIT, but will return home to exercise as they see fit without personalized instruction and coaching. They will be remotely monitored, but will not receive feedback unless any adverse events are noted
  Interventions: Other: Comparator

INTERVENTIONS:
Behavioral: REmotely Monitored, Mhealth (REMM) supported High Intensity Interval Training (HIIT) — REmotely Monitored, Mhealth (REMM) supported High Intensity Interval Training (HIIT) The intervention consists of high intensity interval training, consisting of a 30-minute exercise session that includes 10 x 1-minute intervals of high intensity 3x/week (e.g., Monday, Wednesday, Friday) and supplemented with 2 sessions per week of strength, balance, and mobility exercises (e.g., Tuesday, Thursday). Exercise will be supported by an activity tracker, which will allow study personnel to track patient heart rates during exercise on a daily basis, allowing them to provide individualized feedback and coaching.
  Arms: REmotely Monitored, Mhealth (REMM) supported High Intensity Interval Training (HIIT)
Other: Comparator — Patients randomized to the control arm will receive the same technology platform and education on exercise options, including HIIT, but will return home to exercise as they see fit without personalized instruction and coaching. They will be remotely monitored, but will not receive feedback unless any adverse events are noted
  Arms: Comparator

SUMMARY:
REmotely Monitored, Mobile Health-Supported High Intensity Interval Training after COVID-19 critical illness (REMM-HIIT-COVID-19)

DETAILED DESCRIPTION:
REmotely Monitored, Mhealth (REMM) supported High Intensity Interval Training (HIIT to improve recovery after Intensive Care Unit (ICU) discharge in patients with COVID-19 (REMM-HIIT-ICU-COVID) will evaluate the feasibility of clinical-, physiological- and patient-centered outcomes associated with a remotely monitored, Mhealth-supported high intensity interval rehabilitation exercise training to improve the functional recovery of survivors who have experienced critical illness with COVID-19 and have been discharged home from the hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years
2. ICU admission and subsequent discharge for primary diagnosis of COVID-19 respiratory failure or infection requiring intubation and mechanical ventilation for > 48 hours with an ICU length of stay of ≥ 4 days.
3. Ability to ambulate with or without a gait aid prior to hospital discharge
4. Expected hospital discharge directly back to patient's residence (not to a skilled nursing facility, inpatient rehabilitation center, or long-term acute care hospital)

Exclusion Criteria:

1. Not ambulating independently prior to COVID-19 illness (use of a gait aid permitted)
2. Functional impairment resulting in inability to exercise at hospital discharge (including need for home oxygen requirement)
3. Unable or unwilling to follow coaching via mobile-health iPhone interaction
4. Any absolute contraindications to exercise (as outlined in the American Thoracic Society Guidelines for Cardiopulmonary Exercise Testing), including but not limited to:

   1. Recent (< 5 days) acute primary cardiac event
   2. Unstable Angina
   3. Uncontrolled dysrhythmias causing symptoms or hemodynamic compromise
   4. Symptomatic aortic stenosis
   5. Uncontrolled symptomatic heart failure
   6. Acute myocarditis or pericarditis
   7. Suspected or known dissecting aneurysm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Peak oxygen consumption (V02P) at 3 months after hospital discharge | 3 months post-discharge

SECONDARY OUTCOMES:
Change in 6 minute walk test distance from baseline to 3 months after hospital discharge | Hospital discharge (baseline), 3 months post-discharge
  distance walked in 6 minutes
Change in muscle mass from baseline to 3 months after hospital discharge | Hospital discharge (baseline), 3 months post-discharge
  Measured by muscle sound
Change in muscle strength from baseline to 3 months after hospital discharge | Hospital discharge (baseline), 3 months post-discharge
  Measured by Fried Frailty (includes Hand Grip strength)
Change in muscle strength from baseline to 3 months after hospital discharge | Hospital discharge (baseline), 3 months post-discharge
  Measured by quadriceps strength (Quadricep muscle dynamometry)
Cognition at 3 months after hospital discharge | 3 months post-discharge
  Measured by Repeatable Battery for Assessment of Neuropsychological Status (RBANS)
Change in cognition from baseline to 3 months after hospital discharge. | Hospital discharge (baseline), 3 months post-discharge
  Measured by Montreal Cognitive Assessment (MOCA)
Change in cognition from baseline to 3 months after hospital discharge. | Hospital discharge (baseline), 3 months post-discharge
  Measured by Hayling Sentence Completion
Change in cognition from baseline to 3 months after hospital discharge. | Hospital discharge (baseline), 3 months post-discharge
  Measured by PROMIS Cognitive function
Change in cognition from 3 months to 6 months after hospital discharge. | 3 months post-discharge, 6 months post-hospital discharge
  Measured by PROMIS Cognitive function
Change in quality of life from baseline to 3 months after hospital discharge. | Hospital discharge (baseline), 3 months post-discharge
  Measured by Sociodemographic survey
Change in quality of life from baseline to 3 months after hospital discharge. | Hospital discharge (baseline), 3 months post-discharge
  Measured by Employment Survey
Change in quality of life from baseline to 3 months after hospital discharge. | Hospital discharge (baseline), 3 months post-discharge
  Measured by EQ-5D-5L
Change in quality of life from baseline to 3 months after hospital discharge. | Hospital discharge (baseline), 3 months post-discharge
  Measured by Katz ADL/ Lawton IADL
Change in quality of life from baseline to 3 months to 6 months after hospital discharge. | 3 months post-discharge, 6 months post-hospital discharge
  Measured by Sociodemographic Survey
Change in quality of life from baseline to 3 months to 6 months after hospital discharge. | 3 months post-discharge, 6 months post-hospital discharge
  Measured by Employment Survey
Change in quality of life from baseline to 3 months to 6 months after hospital discharge. | 3 months post-discharge, 6 months post-hospital discharge
  Measured by EQ-5D-5L
Change in quality of life from baseline to 3 months to 6 months after hospital discharge. | 3 months post-discharge, 6 months post-hospital discharge
  Measured by Katz ADL/ Lawton IADL

OTHER OUTCOMES:
Change in biomarkers of aging and resilience, and mitochondrial function from baseline to 3 months post-discharge | Hospital discharge (baseline), 3 months post-discharge
  Measured by peripheral blood mononuclear cell (PBMC)
Change in biomarkers of aging and resilience, and mitochondrial function from baseline to 3 months post-discharge | Hospital discharge (baseline), 3 months post-discharge
  Measured by plasma

CONTACTS AND LOCATIONS:
Overall Officials: Paul Wischmeyer, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No